CLINICAL TRIAL: NCT01604850
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Study to Investigate the Efficacy and Safety of GS-7977 + Ribavirin for 12 or 16 Weeks in Treatment Experienced Subjects With Chronic Genotype 2 or 3 HCV Infection
Brief Title: Sofosbuvir + Ribavirin for 12 or 16 Weeks in Treatment Experienced Subjects With Chronic Genotype 2 or 3 HCV Infection (FUSION)
Acronym: FUSION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-334-0108
Record Dates: First submitted 2012-05-21; First posted 2012-05-24 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Hepatitis C
Keywords: HCV genotype 2 (GT-2); HCV genotype 3 (GT-3); HCV; Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy; Treatment Experienced; GS-7977; Ribavirin
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Sofosbuvir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SOF+RBV+placebo (Experimental): Participants were randomized to receive SOF+RBV for 12 weeks followed by placebo to match SOF plus placebo to match RBV for 4 weeks.
  Interventions: Drug: SOF; Drug: RBV; Drug: Placebo to match SOF; Drug: Placebo to match RBV
- SOF+RBV (Experimental): Participants were randomized to receive SOF+RBV for 16 weeks.
  Interventions: Drug: SOF; Drug: RBV

INTERVENTIONS:
Drug: SOF — Sofosbuvir (SOF) 400 mg tablet was administered orally once daily.
  Other Names: Sovaldi®; GS-7977; PSI-7977
Drug: RBV — Ribavirin (RBV) tablets was administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg).
Drug: Placebo to match SOF — Placebo to match SOF was administered orally once daily.
  Arms: SOF+RBV+placebo
Drug: Placebo to match RBV — Placebo to match RBV was administered orally twice daily.
  Arms: SOF+RBV+placebo

SUMMARY:
This study was to assess the safety and efficacy of sofosbuvir in combination with ribavirin (RBV) administered for 12 or 16 weeks in participants with genotypes 2 or 3 hepatitis C virus (HCV) infection as assessed by the proportion of participants with sustained virologic response (SVR) 12 weeks after discontinuation of therapy (SVR12).

ELIGIBILITY:
Inclusion Criteria:

* Infection with HCV genotype 2 or 3
* Had cirrhosis determination
* Prior treatment failure
* Screening laboratory values within defined thresholds
* Subject had not been treated with any investigational drug or device within 30 days of the screening visit
* Use of highly effective contraception methods if female of childbearing potential or sexually active male

Exclusion Criteria:

* Prior exposure to an direct-acting antiviral targeting the HCV nonstructural protein (NS)5B polymerase
* Pregnant or nursing female or male with pregnant female partner
* Current or prior history of clinical hepatic decompensation
* History of clinically significant illness or any other major medical disorder that may have interfered with subject treatment, assessment or compliance with the protocol
* Excessive alcohol ingestion or significant drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (66):
- United States (51):
  - SCTI Research Foundation, Coronado, California
  - Kaiser Permanente, Los Angeles, California
  - Peter J. Ruane, MD, Inc., Los Angeles, California
  - Anthony Mills MD, Inc., Los Angeles, California
  - UCSD Antiviral Research Center, San Diego, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Kaiser Permanente, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - South Denver Gastroenterology, PC, Englewood, Colorado
  - Whitman Walker Clinic, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Borland-Groover Clinic Baptist, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Advanced Research Institute, New Port Richey, Florida
  - Orlando Immunology Center (ACH), Orlando, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - South Florida Center of Gastroenterology, P.A., Wellington, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - Graves-Gilbert Clinic, Bowling Green, Kentucky
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Johns Hopkins University, Lutherville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - Henry Ford Health System, Novi, Michigan
  - Minnesota Gastroenterology, P.A., Minneapolis, Minnesota
  - Kansas City Gastroenterology and Hepatology, Kansas City, Missouri
  - Comprehensive Clinical Research, Berlin, New Jersey
  - ID Care, Hillsborough, New Jersey
  - Southwest C.A.R.E. Center, Santa Fe, New Mexico
  - Binghamton Gastroenterology Associates, Binghamton, New York
  - Mount Sinai School of Medicine, New York, New York
  - Asheville Gastroenterology Associates, P.A., Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Gastro One, Germantown, Tennessee
  - Nashville Gastrointestinal Specialists, Inc, Nashville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Southwest Infectious Disease Clinical Research, Inc., Dallas, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Metropolitan Research, Fairfax, Virginia
  - Inova Fairfax Hospital Center for Liver Diseases, Falls Church, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Bon Secours St. Mary's Hospital of Richmond, Inc., Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Canada (11):
  - University of Calgary, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Gordon & Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - University of British Columbia, Vancouver, British Columbia
  - (G.I.R.I.) Gastrointestinal Research Institute, Vancouver, British Columbia
  - University of Manitoba Health Sciences Center, Winnipeg, Manitoba
  - The Ottawa Hospital, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Hopital St. Luc, Montreal, Quebec
- New Zealand (2):
  - Auckland Clinical Studies Limited, Auckland
  - Christchurch Hospital, Christchurch
- Puerto Rico (2):
  - Clinical Research Puerto Rico Inc, San Juan, PR
  - Fundacion De Investigacion De Diego, San Juan, PR

REFERENCES:
- [Derived] Younossi ZM, Stepanova M, Sulkowski M, Naggie S, Puoti M, Orkin C, Hunt SL. Sofosbuvir and Ribavirin for Treatment of Chronic Hepatitis C in Patients Coinfected With Hepatitis C Virus and HIV: The Impact on Patient-Reported Outcomes. J Infect Dis. 2015 Aug 1;212(3):367-77. doi: 10.1093/infdis/jiv005. Epub 2015 Jan 12. PMID 25583164
- [Derived] Stepanova M, Nader F, Cure S, Bourhis F, Hunt S, Younossi ZM. Patients' preferences and health utility assessment with SF-6D and EQ-5D in patients with chronic hepatitis C treated with sofosbuvir regimens. Aliment Pharmacol Ther. 2014 Sep;40(6):676-85. doi: 10.1111/apt.12880. Epub 2014 Jul 15. PMID 25040192
- [Derived] Jacobson IM, Gordon SC, Kowdley KV, Yoshida EM, Rodriguez-Torres M, Sulkowski MS, Shiffman ML, Lawitz E, Everson G, Bennett M, Schiff E, Al-Assi MT, Subramanian GM, An D, Lin M, McNally J, Brainard D, Symonds WT, McHutchison JG, Patel K, Feld J, Pianko S, Nelson DR; POSITRON Study; FUSION Study. Sofosbuvir for hepatitis C genotype 2 or 3 in patients without treatment options. N Engl J Med. 2013 May 16;368(20):1867-77. doi: 10.1056/NEJMoa1214854. Epub 2013 Apr 23. PMID 23607593

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in a total of 57 study sites in the United States, Canada, and New Zealand. The first participant was screened on 04 June 2012. The last participant observation was on 08 May 2013.
Pre-assignment Details: 277 participants were screened and 202 were randomized. Of those participants randomized, 201 received at least one dose of study drug, and comprise the Safety Analysis Set; 195 of those participants with genotypes 2 or 3 HCV infection were treated and comprise the Full Analysis Set.
Groups:
- SOF+RBV+Placebo: Participants were randomized to receive sofosbuvir (SOF)+ribavirin (RBV) for 12 weeks, followed by placebo to match sofosbuvir plus placebo to match RBV for 4 weeks.
  Sofosbuvir (400 mg) was administered as an oral tablet and RBV (1000-1200 mg) as 200 mg oral tablets. Placebo to match sofosbuvir and placebo to match RBV were also administered as oral tablets.
- SOF+RBV: Participants were randomized to receive sofosbuvir+RBV for 16 weeks.
  Sofosbuvir (400 mg) was administered as an oral tablet and RBV (1000-1200 mg) as 200 mg oral tablets.
Period: Overall Study
Arm/Group | SOF+RBV+Placebo | SOF+RBV
Started | 103 | 99
Enrolled and Treated | 103 | 98
Completed | 51 | 69
Not Completed | 52 | 30
Not completed — Enrolled but never treated | 0 | 1
Not completed — Efficacy Failure | 50 | 29
Not completed — Lost to Follow-up | 1 | 0
Not completed — Subject withdrew consent | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants in the Safety Analysis Set (randomized and received at least 1 dose of study drug) were analyzed for baseline characteristics.
Groups:
- SOF+RBV+Placebo: Participants were randomized to receive sofosbuvir+RBV for 12 weeks, followed by placebo to match sofosbuvir plus placebo to match RBV for 4 weeks.
  Sofosbuvir (400 mg) was administered as an oral tablet and RBV (1000-1200 mg) as 200 mg oral tablets. Placebo to match sofosbuvir and placebo to match RBV were also administered as oral tablets.
- Total: Total of all reporting groups
Arm/Group | SOF+RBV+Placebo | SOF+RBV | Total
Number analyzed (Participants) | 103 | 98 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (7.7) | 54 (7.8) | 54 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 61
  Male | 73 | 67 | 140
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 5 | 1 | 6
  White | 88 | 86 | 174
  Asian | 7 | 5 | 12
  American Indian/ Alaska Native/ First Nations | 1 | 3 | 4
  Hawaiian or Pacific Islander | 0 | 1 | 1
  Other | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 74 | 76 | 150
  Canada | 26 | 17 | 43
  New Zealand | 3 | 5 | 8
Hepatitis C Virus (HCV) genotype [Number; unit: participants]
  Genotype 1 | 3 | 3 | 6
  Genotype 2 | 36 | 32 | 68
  Genotype 3 | 64 | 63 | 127
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.5 (0.67) | 6.5 (0.63) | 6.5 (0.65)
HCV RNA Category [Number; unit: participants]
  < 6 log10 IU/mL | 26 | 29 | 55
  ≥ 6 log10 IU/mL | 77 | 69 | 146
IL28 Genotype [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 31 | 30 | 61
    CT | 53 | 56 | 109
    TT | 19 | 12 | 31
Cirrhosis (Y/N) [Number; unit: participants]
  No | 66 | 66 | 132
  Yes | 36 | 32 | 68
  Missing | 1 | 0 | 1
Response to Prior HCV Treatment [Number; unit: participants]
  Nonresponse | 25 | 25 | 50
  Relapse/Breakthrough | 78 | 73 | 151

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving SVR12
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ, ie, < 25 IU/mL) 12 weeks after cessation of therapy.
  For the purposes of this efficacy analysis, the posttreatment period began after the end of active treatment (following Week 12 for the SOF+RBV+placebo arm, and Week 16 for the SOF+RBV arm).
Time Frame: Posttreatment Week 12
Population: The Full Analysis Set included all participants with genotype 2 or 3 HCV infection who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV+Placebo | SOF+RBV
Number analyzed (Participants) | 100 | 95
percentage of participants | 51.0 | 72.6
Statistical Analysis 1: Comparison: SOF+RBV+Placebo vs SOF+RBV; A sample size of 100 subjects in each group would provide over 97% power to detect at least 20% improvement in SVR12 rate from the assumed null rate of 25% using 2-sided exact 1-sample binomial test at significance level of 0.025; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — P-value is from the Cochran-Mantel-Haenszel (CMH) test stratified by the randomization stratification factor (ie, presence/absence of cirrhosis, genotype 2 or 3); Proportion difference = -22.4, 95% CI 2-sided [-34.4 to -10.3] — The difference in proportions between treatment groups and associated 95% confidence interval (CI) are calculated based on stratum-adjusted Mantel-Haenszel proportions

2. Primary Outcome: Adverse Events Leading to Permanent Discontinuation of Study Drug
Description: Adverse events which led to permanent discontinuation of study drug may or may not have been related to study treatment.
Time Frame: Baseline to Week 16
Population: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | SOF+RBV+Placebo | SOF+RBV
Number analyzed (Participants) | 103 | 98
participants | 1 | 0

3. Secondary Outcome: Percentage of Participants Achieving SVR4
Description: SVR4 was defined as HCV RNA < LLOQ 4 weeks after cessation of therapy.
  For the purposes of this efficacy analysis, the posttreatment period began after the end of active treatment (following Week 12 for the SOF+RBV+placebo arm, and Week 16 for the SOF+RBV arm).
Time Frame: Posttreatment Week 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV+Placebo | SOF+RBV
Number analyzed (Participants) | 100 | 95
percentage of participants | 56.0 | 76.8

4. Secondary Outcome: Percentage of Participants Achieving SVR24
Description: SVR24 was defined as HCV RNA < LLOQ 24 weeks after cessation of therapy.
  For the purposes of this efficacy analysis, the posttreatment period began after the end of active treatment (following Week 12 for the SOF+RBV+placebo arm, and Week 16 for the SOF+RBV arm).
Time Frame: Posttreatment Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV+Placebo | SOF+RBV
Number analyzed (Participants) | 100 | 95
percentage of participants | 50.0 | 71.6

5. Secondary Outcome: Percentage of Participants With Viral Breakthrough
Description: Viral breakthrough was defined as HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while receiving treatment, confirmed with 2 consecutive values (second confirmation value could be posttreatment), or last available on-treatment measurement with no subsequent follow-up values.
  For the purposes of this efficacy analysis, assessments were made during active treatment (up to Week 12 for the SOF+RBV+placebo arm, and Week 16 for the SOF+RBV arm).
Time Frame: Up to 16 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV+Placebo | SOF+RBV
Number analyzed (Participants) | 100 | 95
percentage of participants | 0.0 | 0.0

6. Secondary Outcome: Percentage of Participants With Viral Relapse
Description: Viral relapse was defined as HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at end of treatment, confirmed with 2 consecutive values or last available posttreatment measurement.
  For the purposes of this efficacy analysis, the posttreatment period began after the end of active treatment (following Week 12 for the SOF+RBV+placebo arm, and Week 16 for the SOF+RBV arm).
Time Frame: End of treatment to posttreatment Week 24
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SOF+RBV+Placebo | SOF+RBV
Number analyzed (Participants) | 100 | 95
participants | 47 | 26

ADVERSE EVENTS:
Time Frame: Baseline to posttreatment Week 24 plus 30 days
Arm/Group | SOF+RBV+Placebo | SOF+RBV
Serious Adverse Events (participants affected / at risk) | 5/103 | 3/98
Other Adverse Events (participants affected / at risk) | 92/103 | 86/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV+Placebo (N=103) | SOF+RBV (N=98)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV+Placebo (N=103) | SOF+RBV (N=98)
Anaemia (Blood and lymphatic system disorders) | 11 | 4
Nausea (Gastrointestinal disorders) | 22 | 20
Diarrhoea (Gastrointestinal disorders) | 15 | 6
Abdominal pain (Gastrointestinal disorders) | 6 | 5
Dyspepsia (Gastrointestinal disorders) | 6 | 3
Constipation (Gastrointestinal disorders) | 2 | 5
Fatigue (General disorders) | 46 | 46
Irritability (General disorders) | 15 | 11
Pain (General disorders) | 4 | 5
Upper respiratory tract infection (Infections and infestations) | 6 | 5
Contusion (Injury, poisoning and procedural complications) | 4 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5
Headache (Nervous system disorders) | 26 | 32
Dizziness (Nervous system disorders) | 6 | 5
Dysgeusia (Nervous system disorders) | 3 | 6
Disturbance in attention (Nervous system disorders) | 6 | 1
Insomnia (Psychiatric disorders) | 21 | 28
Anxiety (Psychiatric disorders) | 8 | 9
Depression (Psychiatric disorders) | 6 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 7
Rash (Skin and subcutaneous tissue disorders) | 7 | 12
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 5
Decreased Appetite (Metabolism and nutrition disorders) | 9 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years